CLINICAL TRIAL: NCT04245527
Title: Joovvin' for Hormonal Health
Brief Title: Use of Infrared Photomodulation for Hormonal Balance (Joovvin' for Hormonal Health)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ProofPilot (Industry)
Collaborators: Joovv (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2216
Record Dates: First submitted 2020-01-25; First posted 2020-01-29 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Testosterone Deficiency; Estrogen Deficiency

STUDY DESIGN:
Intervention Model Description: Enrolled individuals will receive a Joovv solo for the 8 week study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Study Arm (Experimental): 20 minutes Joovv Solo every day for 8 weeks.
  Interventions: Device: Joovv Infrared Light Device

INTERVENTIONS:
Device: Joovv Infrared Light Device — Joovv is the leading manufacturer of personal, in-home red light therapy devices

SUMMARY:
8-week pilot study looking at the impact of Joovv's infrared photo modulation product on male and female hormone levels.

ELIGIBILITY:
Inclusion Criteria:

* United States resident

Exclusion Criteria:

* current Joovv or other photomodulation therapy user
* under medical supervision for medically treatable illness
* significant travel during study period
* use of birth control

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-01-31 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Testosterone Change | baseline to week 8
  in males, change from baseline to week 8
change of thyroid-stimulating hormone (TSH) | baseline to week 8
  in females change in estrogen and progesterone from baseline to week 8
Self report general wellness | baseline to week 8
  series of questions at baseline and week 8 on general wellness (modified Short Form-36)

CONTACTS AND LOCATIONS:
Locations (1):
- ProofPilot (Virtual Study: https://p.proofpilot.com), New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
there is no current plan to make IPD available to other researchers